CLINICAL TRIAL: NCT03231215
Title: The Effect of Adding Dexamethasone to Epidural Bupivacaine for Total Knee Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed galal aly, Assistant Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17100211
Record Dates: First submitted 2017-07-25; First posted 2017-07-27 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- controlled group (Placebo Comparator): Group І (control group): the patients received 15 ml epidural plain bupivacaine (0.5%) +2 ml normal saline Group (BS).
  Interventions: Drug: Dexamethasone
- dexamethasone group (Active Comparator): Group II (dexamethasone group):- the patients received 15 ml epidural plain bupivacaine (0.5%) + 8mg dexamethasone (2ml) Group (BD)
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — dexamethasone + plain Bupivacaine injected epidurally.
  Other Names: Decadrone

SUMMARY:
The purpose of this study was to evaluate the efficacy of dexamethasone when added to epidural bupivacaine on the duration of postoperative analgesia in patients underwent total knee replacement surgery.

DETAILED DESCRIPTION:
Fifty patients underwent total knee replacement were included in the study. The patients (11 male and 39 female) were classified into two equal groups:- The patients received 15 mL plain bupivacaine + 2 mL (BS), or 8 mg dexamethasone (BD). The total volume injected in both groups was 17 ml.

Postoperative records:

1. Pain score (NRS) at base line, then every 4 hrs for 24 hrs.
2. Frequency of rescue analgesia.
3. Postoperative side effects like nausea, vomiting, and over sedation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for total knee replacement surgery.
2. ASA Physical status I,II,III.

Exclusion Criteria

1. Patients' refusal.
2. Uncooperative patients / Not able to understand pain assessment test.
3. Patients with history of allergy to the used drugs.
4. Significant liver disease.
5. Pregnancy.
6. Any contraindication for epidural anesthesia
7. Failed technique.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-07-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
duration of postoperative analgesia (NRS) | 24 hrs postoperative
  first patient request for analgesia or NRS 4 or more